CLINICAL TRIAL: NCT05703139
Title: Efficacy of the Triangle Operation on Clinical Outcomes in Patients With Pancreatic Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Hossam Abdellatif Mohamed, assistant lecturer, Sohag University
Other Study IDs: Soh-Med-23-01-15
Record Dates: First submitted 2023-01-16; First posted 2023-01-27 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Hepato-Biliary Precancerous Condition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: TRIANGLE procedure — The Triangle procedure aims to develop a novel method for patients with locally advanced pancreatic cancer after neoadjuvant therapy and was described in 2017. The basis of this operation is the notice that after neoadjuvant therapy conventional imaging fails to differentiate between actual tumor encasement and only fibrotic residual tissue mainly to the arterial structures

SUMMARY:
We aimed to analyze postoperative short-and long-terms clinical outcomes after the Triangle procedure in patients with Pancreatic head, periampullary and duodenal cancer.

DETAILED DESCRIPTION:
After laparotomy and exploration of the abdominal cavity to rule out peritoneal or hepatic metastases, the initial steps of the operation were to determine if there was true arterial tumor infiltration, along the Celiac Artery, Hepatic Artery or Superior Mesenteric Artery. To clarify this, an "arteryfirst" maneuver was performed. The strategy depended on the results of preoperative imaging defining the site of the most likely tumor infiltration. The SMA was approached from a left-sided infracolic approach if tumors of the body or tail of the pancreas were suspected to infiltrate the artery from this direction or from a posterior approach in respective situations. Once the arterial level of suspected attachment/encasement was reached, a frozen section was performed to confirm or exclude viable tumor tissue at this site. In case of remaining viable tumor, most patients will not qualify for further surgical therapy at this point. In contrast, if frozen section confirms fibrous tissue without viable tumor, this offers the possibility to perform a radical but artery-sparing procedure, All other surgical steps are carried out as usual during partial pancreatoduodenectomy (PD), distal (DP) or total pancreatectomy. Anatomic TRIANGLE bordered by the SMA, CA and PV confirming the complete removal of all soft tissue usually contained within these borders.

ELIGIBILITY:
Inclusion Criteria:

* No age restriction or Gender exclusion, all diagnosed fit patients with pancreatic head, periampullary and duodenal cancer will be included.

Exclusion Criteria:

* Unfit or inoperable patients will be excluded.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study includes cases that match our eligibility criteria No age restriction or Gender exclusion, all diagnosed fit patients with pancreatic head, periampullary and duodenal cancer will be included, Unfit or inoperable patients will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-11-21 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy of the Triangle operation on clinical outcomes in patients with Pancreatic Cancer Efficacy of the Triangle operation on clinical outcomes in patients with Pancreatic Cancer | 6 months
  no recurrence observed

SECONDARY OUTCOMES:
Efficacy of the Triangle operation on clinical outcomes in patients with Pancreatic Cancer | 1 year
  This study aims to evaluate postoperative short- and long-terms clinical outcomes after the Triangle procedure in patients with pancreatic head, periampullary and duodenal cancers.
  Operative time will be defined from the time of incision to the closure of the skin.
  Short-term outcome starts from the date of surgery until date of discharge those post-operative complications will be categorized according to the Clavien-Dindo Grading System (Dindo et al., 2004).
  Post-operative pancreatic fistula (POPF) will be defined according to the International Study Group on Pancreatic Fistula (ISGPF) (Bassi et al., 2005).
  Post-operative bile leakage will be defined according to the international study group of liver surgery (ISGLS) (Koch et al., 2011).

CONTACTS AND LOCATIONS:
Overall Officials: asem al mohamed, professor, Study Director — Sohag University; omar ab sayed, professor, Study Chair — Sohag University; emad al ahmed, lecturer, Study Chair — Sohag University
Locations (1):
- Sohag University, Sohag, Nasser City, Egypt

IPD SHARING:
Plan to Share IPD: Undecided